CLINICAL TRIAL: NCT06753981
Title: Efficacy and Safety of Triple-targeted Drug Therapy in Treatment-naive Patients With Non-low-risk PAH: A Real-world, Multicenter Study
Status: Recruiting | Type: Observational
Sponsor: Qianfoshan Hospital (Other)
Collaborators: Chinese Academy of Medical Sciences, Fuwai Hospital (Other); Jianghan University Affiliated Hospital (Unknown)
Responsible Party: Principal Investigator, GuanghaiWang, Dr., Qianfoshan Hospital
Other Study IDs: YXLL-KY-2024 (124)
Record Dates: First submitted 2024-12-22; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Arterial Pulmonary Hypertension (PAH)
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Endothelin Receptor Antagonists

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-low-risk PAH treatment-naive patients
  Interventions: Drug: Endothelin receptor antagonist (ERA) combined with PDE5i/sGC agonist dual therapy prostacyclin drugs

INTERVENTIONS:
Drug: Endothelin receptor antagonist (ERA) combined with PDE5i/sGC agonist dual therapy prostacyclin drugs — Endothelin receptor antagonist (ERA) combined with PDE5i/sGC agonist dual therapy prostacyclin drugs Including macitentan sildenafil/tadalafil or riociguat selexipag/epoprostenol.

SUMMARY:
This study is a multicenter, prospective, observational study aimed at investigating the efficacy and safety of triple targeted drug therapy in patients with arterial pulmonary hypertension (PAH) who are not at low risk and are receiving initial treatment. The prognosis of arterial pulmonary hypertension is explored.

ELIGIBILITY:
Inclusion Criteria:

* Consent and sign the informed consent form
* Non-low-risk PAH treatment-naive patients

Exclusion Criteria:

* Positive acute vascular response test for idiopathic/hereditary/drug-related arterial pulmonary hypertension
* Pulmonary veno-occlusive disease/pulmonary capillary hemangiomatosis (PVOD/PCH) with arterial pulmonary
* Pregnant or lactating women
* Suffering from mental illness or cognitive impairment
* PAH patients with concurrent malignant tumors
* Patients with moderate to severe hepatic impairment, renal impairment, and severe anemia
* Currently participating in other interventional clinical studies
* Key clinical data is incomplete, or the investigator considers that the patient has other factors that make them unsuitable for this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with arterial pulmonary hypertension
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2026-11-14 (Estimated); Study Completion 2027-02-14 (Estimated)

PRIMARY OUTCOMES:
Pulmonary Vascular Resistance (PVR) | Up to 3 months

SECONDARY OUTCOMES:
N terminal pro B type natriuretic peptide （NT-proBNP） | Up to 3 months
6-minute walking distance | Up to 3 months
mean pulmonary arterial pressure (mPAP) | Up to 3 months
cardiac index (CI) | Up to 3 months
WHO Heart Function Classification | Up to 3 months
Oxygen Saturation of Mixed Venose Blood (SvO2) | Up to 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Respiratory, The First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital, #16766, Jingshi Road, Jinan City, Shandong Province, China, Jinan, Shandong, China